CLINICAL TRIAL: NCT02894814
Title: My Health - My Medication. A Controlled Investigation of Patient Involvement in Administration of Medication in Hospitalized Medical Patients
Brief Title: My Health - My Medication. Patient Involvement in Administration of Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Appel, Research Nurse, Central Jutland Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6300002A; 1-16-02-124-16 (Other: the Danish Data Protection Agency)
Record Dates: First submitted 2016-05-30; First posted 2016-09-09 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Medical Patients
Keywords: Self administration; Medication; Inpatient; Self-care; Self-management; Medical patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Basic intervention (Active Comparator): Elements of One-Stop Dispensing (use of own medication, placed in bedside locker, partly or self-administration of medication during hospitalization)
  Interventions: Behavioral: One-Stop Dispensing
- Extended intervention (Active Comparator): Elements of One-Stop Dispensing and focused dialogue with the patients about their medication during the hospitalization.
  Interventions: Behavioral: One-Stop Dispensing and focused dialogue
- Observational part of the study (No Intervention): Data collection on patients under the traditional medication system

INTERVENTIONS:
Behavioral: One-Stop Dispensing — Use of own medication, review of the patient's medication, partly or self-administration of medication during hospitalization under support from the health personnel to improve adherence, knowledge and feeling safe about the medication.
  Arms: Basic intervention
Behavioral: One-Stop Dispensing and focused dialogue — Besides the elements of One-Stop Dispensing focused dialogue about the patient's medicine during hospitalization and at discharge to improve adherence, knowledge and feeling safe about the medication
  Arms: Extended intervention

SUMMARY:
The primary purpose of this study is to investigate if patient involvement in the medication procedures through elements of the medication system One-Stop Dispensing (use of own medication, placed in bedside locker, partly or self-administration of medication) and focused dialogue about medication can maintain or improve the patients' health literacy to perform the prescribed medical treatment during and after hospitalization.

The hypothesis is, that involving the patient in the medication procedure and focused dialogue about the medicine during hospitalization will improve the patients' health literacy measured by patient adherence, patient knowledge and perceptions of safety about the medication. It is further expected that more time will be spent together with the patient, and that the new medication procedures will be cost-neutral.

DETAILED DESCRIPTION:
More people live with chronic diseases and therefore it is important for the healthcare system to develop and organize initiatives that involve patients in their treatment.

In Denmark dispensing and administration of medication during hospitalization is a process where the health staff has completely taken the responsibility from the patient, leaving unused resources among patients and their relatives.

In general non-adherence to medication in patients with chronic medical diseases is a common problem, which contributes to adverse health outcomes, increase healthcare expenditures and reduce quality of life.

One-Stop Dispensing (use of own medication, placed in bedside locker, partly or self-administration of medication during hospitalization), which is a medication system developed in United Kingdom in the 1990s, could be an important part of a shift in the healthcare system toward increasing patient involvement. Use of own medication and self-administration aims, among other things, to increase adherence and the patient's knowledge and understanding of their medication. One-Stop Dispensing has so far only been tested on elective surgical patients in Denmark, which is why this study set out to investigate acute hospitalized medical patients.

To investigate the effect of the medication system One-Stop Dispensing in Danish medical patients the investigators planned a study including two designs. An observational before and after implementing One-Stop Dispensing study and a randomized controlled study for the intervention period.

Enrolment for an observational part of the study will begin in April 2016 with data collection on patients under the traditional medication system.

In October 2016 enrolment will then begin for the intervention period including randomization to a basic intervention including the elements of One-Stop Dispensing or an extended intervention which besides One-Stop Dispensing also include a dialogue with the patients about their medication during the hospitalization and at discharge. The data collection will end in March 2017.

The research team will identify and verify patient eligibility. All participants will need to provide informed written consent. For recruitment and informed consent, project information will be discussed with the participants.

Baseline variables will be collected at admission and in the intervention period prior to randomization. This includes questionnaire and baseline characteristics such as age, sex and diagnosis. The primary measure is adherence measured at baseline and 1 month after discharge. Knowledge of the patients' own medication will assessed by a health professional also at baseline and again at discharge.

The study will end after one month follow up is completed for all the included patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients at Diagnostic Center, Regional Hospital Silkeborg, Denmark ≥ age 18 years, who understand, speak and are able to read Danish.

Exclusion Criteria:

* Patients admitted for elective procedures, where admission is expected to be <24 hours
* Patients with significant cognitive problems (dementia, dying, psychotic etc.)
* Patients who abuse medicine or narcotics.
* Patients who have participated in the project during a previous admission.
* Patients who do not use prescribed medicine.
* Patients admitted in the period monday from 8 a.m. until friday 3 p.m.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in adherence to medical treatment | From baseline (admission) to one month after discharge
  Ability to adhere to medical recommendations in general, assessed by questionnaire at baseline (admission to hospital) and 1 month after discharge.

SECONDARY OUTCOMES:
Patient satisfaction | The day at discharge, after admission of an average of 3 days
  Patient satisfaction regarding medication during hospitalization, assessed by questionnaire at discharge
Time spent per patient | Days admitted, an average of 3 days
  Time spent per patient on preparing and administering the medication, assessed by timing time spent in the medication room and together with the patient.
Cost per patient | Days admitted, an average of 3 days
  Financial cost per patient spent on medication primarily assessed on the cost of supplying patient medicines
Knowledge of own medication | Days admitted, an average of 3 days
  Patient's knowledge of own medication assessed by a health professional at baseline (admission to hospital) and at discharge
Change in patient's perception of security and safety regarding medication | From baseline (admission) to one month after discharge
  Patient's perception of safety and security regarding their own medication and general beliefs about medicines, assessed by questionnaire at baseline (admission and 1 month after discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte W Appel, PhD, Principal Investigator — Diagnostic Centre, Regional Hospital Silkeborg, Denmark
Locations (1):
- Diagnostic Centre, Regional Hospital Silkeborg, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided